CLINICAL TRIAL: NCT05892601
Title: Let me Kiss it Better! Maternal Kisses Are Effective in Alleviating Pain, Anxiety, and Fear in Children During Invasive Procedures: A Randomized Controlled Study
Brief Title: Effect of Maternal Kisses on Pain, Anxiety, and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Emre Ciydem, Assistant Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BandirmaOnyediEylulU-SBF-EÇ-01
Record Dates: First submitted 2023-05-25; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Chin Injury
Keywords: Evidence-Based Nursing; Pain Management; Fear; Anxiety
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized controlled experimental study with a single-blind pretest-posttest control group.
Who Masked: Care Provider
Masking Description: Stratified block randomisation method was used to assign the participants to the intervention and control groups. To prevent bias, randomisation was performed by an unbiased nurse who was not involved in the study. In order to control the imbalances that may arise between the intervention and control groups, stratification (2X2) was made according to gender (girls, boys) and age (5,6,7) and an equal number of children were assigned to each group (blocking). Assignments were made according to a list generated by an online randomisation tool. All participants completed the study process and there was no case loss. The parents of the children who participated in the study were unaware of which group their children were in. Since the applications were carried out by the researcher, researcher blinding could not be performed. Therefore, the study is single blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mother kisses were applied to the experimental group. Kisses were delivered by the mother, free of oral ulcers, with a standard 5-second pressing of both lips on the affected body part followed by an exaggerated puckering sound.
  Interventions: Other: Maternal kisses
- Control (No Intervention): The invasive intervention was performed with the standard method in the control group.

INTERVENTIONS:
Other: Maternal kisses — The parents of the children in the experimental group were informed about the process before the application. The parents were asked to approach their child immediately after the invasive procedure was over, call out "Let me kiss it better" and kiss the child from a point not close to the place where the invasive procedure was applied. Kisses were delivered by the mother, free of oral ulcers, with a standard 5-second pressing of both lips on the affected body part followed by an exaggerated puckering sound. Pain, fear, and anxiety scales were administered to the intervention group at the 1st and 5th minutes after the application. Invasive interventions have been applied by researchers who have been working as nurses in the emergency room for 4 years.
  Arms: Intervention

SUMMARY:
Although the effectiveness of maternal kisses for minor injuries in childhood is traditionally accepted, its effect on invasive procedures has not yet been proven. The aim of this study is to determine the effect of maternal kisses applied to children aged 5-7 years on pain, anxiety, and fear levels during invasive procedures. The population of the pretest-posttest single-blind randomized controlled experimental study consisted of 124 children aged 5-7 years who applied to the pediatric gastroenterology clinic , and the sample consisted of 84 children. A stratified block randomization method was used in the study. The maternal kisses were applied to the experimental group during the invasive procedure, and the standard invasive procedure was applied to the control group. The effect of maternal kisses' on reducing pain, anxiety, and fear in children during invasive procedures is being investigated.

DETAILED DESCRIPTION:
Method

Type of study

The design of this study was a randomised controlled experimental study with a single blind pre-test post-test control group. The study was conducted according to CONSORT guidelines.

Hypotheses H01: Mother's kiss during invasive intervention has no effect on pain.

H11: Mother's kiss during invasive intervention has an effect on pain.

H02: Mother's kiss during invasive intervention has no effect on anxiety.

H12: Mother's kiss during invasive intervention has an effect on anxiety.

H03: Mother's kiss during invasive intervention has no effect on fear.

H13: Mother's kiss during invasive intervention has an effect on fear.

Population and Sample

The population of the study consisted of 124 children aged 5-7 years who applied to a private pediatric gastroenterology clinic for diagnosis and treatment between 11 January 2023 and 5 May 2023, and the sample consisted of 84 children. The minimum sample size was calculated with GPower 3.1 Statistical Software. Since the effect size could not be determined in a similar study, a pilot study was conducted with a total of 10 people, five people per group in the intervention and control groups. Pilot applications were not included in the study afterwards. In line with the data obtained from the pilot study, the effect size calculated using the mean and standard deviation of the fear level scores of the children in the intervention and control groups at the 5th minute was d:0.73. Accordingly, for an effect size of d:0.73, alpha:0.05 and 1-alpha:0.95, the number of people to be sampled within each group was determined as 42 and 84 in total. The study was completed with a total of 84 participants. As a result of the PostHoc power analysis performed after the data were collected, the power of the test was determined as 99.9% with 95% confidence (1-alpha), d=0.97 effect size and n=84 participants. The effect size used in the PostHoc analysis was calculated by using the mean and standard deviation of the fear level scores of the children in the intervention and control groups at the 5th minute.

Application

After obtaining the necessary permissions, the data were collected by the researcher through face-to-face interviews. The eligibility of the children and their parents who were admitted to the pediatric gastroenterology clinic and decided to undergo invasive intervention after examination were evaluated. Then, the verbal consent of the children who volunteered to participate in the study and met the inclusion criteria and the written consent of the mothers were obtained. Stratified randomisation method was used to assign the children to the groups. Then, according to the type of intervention to be applied, the child and the parent were included in the relevant section. Blood collection and observation rooms, where invasive interventions are performed, are separated by a screen for one person and designed to protect privacy. All data collection tools except the pain scale were administered to the children in the intervention and control groups as pretest. Mother's kiss was applied to the intervention group. The control group underwent invasive intervention with the standard method. Before the application, it was checked whether the parents had oral ulcers. The parents of the children in the intervention group were informed about the process before the application. Immediately after the invasive procedure was finished, the parent was asked to approach his/her child and say, "Let me kiss you and make it better" and to kiss his/her child from a point not close to where the invasive procedure was performed. Kisses were delivered by mother, free of oral ulcers, with a standard 5-second pressing of both lips on the affected body part followed by an exaggerated puckering sound. Pain, fear and anxiety scales were re-administered to both groups at the 1st and 5th minutes after the application. Invasive interventions were performed by the researchers who had been working as nurses for 4 years and by the medical doctor. The same procedures were repeated for each child who met the inclusion criteria. The parents of the children in the control group remained in the same environment with their child during the invasive intervention. After the application process was completed, the children in the control group were also provided with the mother's kiss application.

Data Evaluation

The data of the study were evaluated using Statistical Package for Social Sciences (SPSS) (23.0) programme in computer environment. The conformity of the data to normal distribution was evaluated by Shapiro-Wilk tests. Number, percentage, mean, standard deviation were used in data analysis, and chi-square test was used to determine homogeneity in categorical variables. Since the data were normally distributed, repeated measures analysis of variance with Bonferroni correction was used for intra-group comparisons and independent samples t test was used for inter-group comparisons. The significance level was determined as p<0.05.

Ethical Aspects of the Study

The study was conducted in accordance with the principles of the Declaration of Helsinki. Ethics committee permission was obtained from Bandırma Onyedi Eylül University Health Sciences Non-Interventional Research Ethics Committee (Date: 18.10.2022, Number:2022-9). Then, permission was obtained from the clinic where the study would be conducted. Before the data were collected, the children and their parents were informed about the purpose and scope of the study and their verbal consent was obtained by asking whether they agreed to participate in the study, and the written consent of the parents who agreed to participate in the study was obtained through the Informed Voluntary Consent Form. Patient rights and privacy as well as ethical rules were observed throughout the whole process.

ELIGIBILITY:
Inclusion Criteria (Mother)

* Being over 18 years of age
* Speaking Turkish
* Having two lips with which to apply the kiss
* Written informed consent

Exclusion Criteria (Mother)

* Having oral ulcers
* Accused or convicted of child abuse or neglect

Inclusion Criteria (Child)

* Being in the age range of 5-7 years
* Admission to pediatric gastroenterology clinic for diagnosis and treatment
* Stable general condition
* Invasive intervention performed in a single attempt
* Not having visual and hearing problems
* Not having any pain (due to illness, side effects of medication, distension)
* Not having a chronic disease (kidney, diabetes, etc.) that requires frequent invasive intervention
* Being at the level of mental development to answer the questions asked
* Speaking and understanding Turkish easily
* Volunteering to participate in the study

Exclusion Criteria (Child)

* Having a history of epilepsy, vertigo and neurological diseases
* History of syncope during blood collection
* Having a disease that causes chronic pain
* Complications during invasive intervention (allergy, syncope, etc.)
* Being in life-threatening condition and taken to the resuscitation room
* Deciding that the child is a forensic case after the examination
* In the intervention group, the parent makes an intervention other than kissing the child within 5 minutes
* In the control group, the parent makes any intervention to his/her child within 5 minutes

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Groups were assigned according to biological sex.
Enrollment: 84 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale | 5th minute
  Wong-Baker Faces Pain Rating Scale: There are 6 different facial expressions scored between 0 and 5 on the scale. A smiling face means no pain, a crying face means unbearable pain. Explain the meaning of facial expressions to the child. Then, they are asked to show the face that best expresses the level of pain when asked. The number on the facial expression specified by the child is recorded. As the score obtained from the scale increases, pain tolerance decreases.

SECONDARY OUTCOMES:
Child Anxiety Scale-State | 5th minute
  Child Anxiety Scale-State (CAS-D):CAS-D is shaped like a thermometer with a light bulb at the bottom and horizontal lines at intervals going upwards. The scale can be used for children over the age of four. To determine the child's anxiety level, say, "Imagine that all your anxious or nervous emotions are on the bulb or the bottom of the thermometer. If you are a little worried or nervous, the emotions may go up a little on the thermometer. If you are very, very worried or nervous, the emotions can run high. How worried is the thermometer or put a line to show that he is angry". To measure state anxiety, the child is asked to mark how he or she is currently feeling. Marked with a transparent meter is placed, then ½ point increase is rounded to the nearest number The possible scores range from 0 to 10.
Child Fear Scale | 5th minute
  Child Fear Scale (CDS): The validity index of the scale was found to be 0.89. The visual structure of the scale makes it easy to use. The CLS includes five distinct facial expressions, ranging from neutral (0=no fear) to frightened (4=severe fear). The scale is scored between 0-4. It can be used by families and/or researchers to evaluate fear before and during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ciydem, Ph.D., Principal Investigator — Bandırma Onyedi Eylül University
Locations (1):
- Uzm. Dr. Engin Demir Muayenehanesi, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No